CLINICAL TRIAL: NCT00440453
Title: Feeding the Patient at Nutritional Risk: Does the Clinical Outcome Improve?
Acronym: EMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Dr. med. Zeno Sanga, University Hospital Inselspital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EMS_CH_2007
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Malnutrition
Keywords: Internal medicine patients
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Normal hospital food
- 2 (Experimental): Nutritional treatment
  Interventions: Other: Nutritional therapy

INTERVENTIONS:
Other: Nutritional therapy — Nutritional therapy by dietician
  Arms: 2

SUMMARY:
The aim of the present study is to take stronger action in solving the problems of malnutrition in the hospital setting and in the first two months after patient's discharge. The main objective is to evaluate the clinical benefit (eg. QoL, body composition and body function) of nutritional intervention (nutritional therapy) in a sample of patients at nutritional risk according to the NRS 2002.

ELIGIBILITY:
Inclusion Criteria:

* all patients coming on station

Exclusion Criteria:

* patients with a screening total score <3 according to the NRS-2002 system
* less than 18 years of age, expected hospital stay less than 4 days
* expected survival less than 1 month
* pregnant or lactating women
* patients with psychiatric disorders
* patients with cardiac failure as defined by the Goldmann classification class >II (recent rest pain, unstable angina pectoris)
* patients with respiratory failure (Peak Flow Rate: PEFR <50%)
* patients with hepatic dysfunction (Child >A)
* patients suffering from an intestinal obstruction or ileus
* patients with renal failure (creatinine >250 μmol/l) or receiving haemodialysis
* patients that are already receiving, or are planned to receive parenteral nutrition
* patients unable to understand the German language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Length of stay | after stay

SECONDARY OUTCOMES:
Quality of life | 2 months after stay
Changes in body weight (measured day 1-2, 8, 28 and 56) and body composition (BMI, MAC, TSF) (measured day 1-2 and 8) | during stay
Changes in muscle function (handgrip dynamometry) (measured day 1-2 and 8) | during stay
Rate of accurately defined complications (infectious and non-infectious) (Table 2). Infectious are defined according to the US Centre of Disease Control [115]. | during stay
Rate of accurately defined post-discharge complications (infectious and non-infectious) (Table 2) | after stay
Rate of re-hospitalization (within 8 weeks after randomisation) | after stay
Rate of mortality | during and after stay

CONTACTS AND LOCATIONS:
Overall Officials: Samuel W Iff, MD, Principal Investigator — University hospital Berne
Locations (1):
- University hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Allison SP. Malnutrition, disease, and outcome. Nutrition. 2000 Jul-Aug;16(7-8):590-3. doi: 10.1016/s0899-9007(00)00368-3. No abstract available. PMID 10906565